CLINICAL TRIAL: NCT03370081
Title: Effects of Capnometry Monitoring in Post Anesthesia Care Unit
Acronym: CAPNOSSPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Principal Investigator, Karine Nouette-Gaulain, M.D; PH.D. Head of department, Anesthesiology and ICU, clinical professor, University Hospital, Bordeaux
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CHUBX2017/18
Record Dates: First submitted 2017-12-04; First posted 2017-12-12 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: VENTILATION; Capnography
Keywords: Capnometry; Capnography; ETCO2; Recovery room; Post-anesthesia care unit
MeSH Terms: conditions — Respiratory Aspiration | interventions — Capnography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAPNO+ (Experimental): END TIDAL CO2(EtCO2) is monitoring and PACU nurses can see the values delivered by the capnography device
  Interventions: Device: CAPNOGRAPHY
- CAPNO- (No Intervention): END TIDAL CO2(EtCO2) is monitoring but PACU nurses cannot see the values delivered by the capnography device

INTERVENTIONS:
Device: CAPNOGRAPHY — MONITORING OF CAPNOMETRY USING ETCO2 METHOD
  Arms: CAPNO+

SUMMARY:
There is few information about the best capnometry value in recovery room for intubated awakening patients. Furthermore, capnometry values could influence ventilation applied by nurses on these patients. The aim of this study is to observe the effects of capnometry monitoring on intubated awakening patients in recovery room.

DETAILED DESCRIPTION:
In France, there is actually no recommandation about capnography monitoring in recovery rooms. Nevertheless, some patients are still ventilated in post-anesthesia care units during awakening period. Alveolar hypoventilation could induce moderate hypercapnia, thereby stimulate central ventilatory command. However, this hypoventilation could delay the clearance of anesthetic gases. Capnometry monitoring could influence ventilation applied to these patients. Recovery rooms nurses would perform moderate hyperventilation in response to hign capnometry values. This method could enhance gases elimination, with faster spontaneous breathing recovery and extubation. Length of stay in recovery room could also be shortened. An objective surrogate of ventilation is maximal End Tidal CO2, if there is no alveolo-capillary gradient abnormality (Obesity, Chronic respiratory disease, Cyanogenic heart disease). Thus, this study will compare the percentage of patients who reached a maximum End Tidal CO2 greater than 45mmHg during awakening period in post-anesthesia care unit (PACU) in 2 groups :

* first group ("non-blind group") with capnography monitoring see by the PACU nurses
* second group ("blind group") with capnography monitoring but PACU nurses cannot see the values Other parameters like the time between ventilator's disconnection and the first ventilatory cycle in spontaneous ventilation, the time between ventilator's disconnection and tracheal extubation or laryngeal mask's withdrawal, the minimal SpO2 reached after tracheal extubation or laryngeal mask withdrawal or the length of stay in PACU are also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Major patients with given written consent
* General anesthesia, induction with Propofol infusion and Target-Controlled Infusion (TCI) remifentanil, relayed with inhaled sevoflurane and TCI remifentanil
* Upper airway control with naso-orotracheal tube or laryngeal mask
* Ventilated normotherm patients in PACU

Exclusion Criteria:

* Minor or pregnant patients
* Obesity with Body Mass Index > 40 kg/m²
* Chronic respiratory disease with SpO2<90% in ambiant air
* Cyanogenic heart disease
* Patients under myorelaxant in PACU

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
End Tidal CO2 up | through awakening period in PACU, an average of 30 minutes
  Percentage of patients who reached a maximum End Tidal CO2 greater than 45mmHg during awakening period in post-anesthesia care unit (PACU)

SECONDARY OUTCOMES:
End Tidal CO2 max 1 | through awakening period in PACU, an average of 15 minutes
  Maximum EtCO2 reached before the first ventilatory cycle in spontaneaous ventilation
End Tidal CO2 max 2 | through awakening period in PACU, an average of 30 minutes
  Maximum EtCO2 reached after the first ventilatory cycle in spontaneous ventilation
respiratory rate | through awakening period in PACU, an average of 15 minutes
  Respiratory rate applied by PACU nurse before the first ventilatory cycle in spontaneous ventilation
spontaneous ventilation time | through awakening period in PACU, an average of 15 minutes
  Time (in minutes) between ventilator's disconnection and the first ventilatory cycle in spontaneous ventilation
time for removal of airway device | through awakening period in PACU, an average of 30 minutes
  Time (in minutes) between ventilator's disconnection and tracheal extubation or laryngeal mask's withdrawal
Spo2 min | through awakening period in PACU, an average of 2 hours
  Minimal SpO2 after tracheal extubation or laryngeal mask withdrawal
length of stay in PACU | through awakening period in PACU, an average of 2 hours
  Length of stay in PACU in minutes
time for oxygenotherapy removal | through awakening period in PACU, an average of 1 hour
  Time (in minutes) between tracheal extubation or laryngeal mask withdrawal and oxygenotherapy weaning

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier Universitaire de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Potvin J, Etchebarne I, Soubiron L, Biais M, Roullet S, Nouette-Gaulain K. Effects of capnometry monitoring during recovery in the post-anaesthesia care unit: a randomized controlled trial in adults (CAPNOSSPI). J Clin Monit Comput. 2022 Apr;36(2):379-385. doi: 10.1007/s10877-021-00661-9. Epub 2021 Feb 7. PMID 33550546